CLINICAL TRIAL: NCT07092839
Title: Investigation of the Plasticity of Deep Brain Structures in Mild Cognitive Impairment and Healthy Aging (PlasMA)
Brief Title: Non-invasive Deep Brain Stimulation to Enhance Motor Skill Acquisition in Individuals With Mild Cognitive Impairment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Friedhelm Hummel (Other)
Collaborators: Clinique Romande de Readaptation (Network); HUG University hospital (Unknown); SNSF (Unknown); The Novartis Foundation (Other); Wyss Center for Bio and Neuroengineering (Other); Fondation Bertarelli (Unknown)
Responsible Party: Sponsor-Investigator, Friedhelm Hummel, Prof. Dr. med., Ecole Polytechnique Fédérale de Lausanne
Organization: Ecole Polytechnique Fédérale de Lausanne (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 2020-00127-wp5m
Record Dates: First submitted 2025-07-10; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Mild Cognitive Impairment (MCI)
Keywords: non-invasive brain stimulation; deep brain stimulation; subcortical; memory; neuro-imaging; transcranial temporal interference stimulation; motor learning
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active stimulation (Experimental): Patterned stimulation (intermittent theta-burst) generating temporal interference in the striatum; see Wessel et al., 2023, Nat Neurosci. for details
  Interventions: Other: transcranial electric stimulation
- Placebo stimulation (Placebo Comparator): Sham stimulation : ramp-up [5 s] immediately followed by ramp-down [5 s] of high-frequency currents (see Vassiliadis et al., 2023, Nat Hum Behav for more details)
  Interventions: Other: transcranial electric stimulation

INTERVENTIONS:
Other: transcranial electric stimulation — tTIS is an innovative non-invasive brain stimulation approach, in which two or more independent stimulation channels deliver high-frequency currents in the kHz range (oscillating at f1 and f1 + Δf). These high-frequency currents are assumed to be too high to effectively modulate neuronal activity. Still, by applying a small shift in frequency, they result in a modulated electric field with the envelope oscillating at the low-frequency Δf (target frequency) where the two currents overlap. The peak of the modulated envelope amplitude can be steered towards specific areas located deep in the brain, by tuning the positions of the electrodes and the current ratio across stimulation channels. Here, we applied tTIS via surface electrodes applying a low-intensity (2mA baseline to peak), sub-threshold protocol following the safety guidelines for low-intensity transcranial electric stimulation in humans.

SUMMARY:
The goal of this study is to investigate the impact of non-invasive deep brain stimulation on motor skill acquisition in individuals with Mild Cognitive Impairment. Participants performed a motor task with non-invasive deep brain stimulation applied to the striatum, which is crucial for motor skill acquisition. The study compared motor skill performance between with the active stimulation and the control stimulation.

DETAILED DESCRIPTION:
This study implemented a randomized, double-blinded, and sham-controlled design, investigating the effects of non-invasive deep brain stimulation on motor skill acquisition in individuals Mild Cognitive Impairment.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Clinical diagnosis of MCI

Exclusion Criteria:

* Unable to consent
* Severe neuropsychiatric (e.g., major depression, severe dementia) or unstable systemic diseases (e.g., severe progressive and unstable cancer, life threatening infectious diseases)
* Severe sensory or cognitive impairment or musculoskeletal dysfunctions prohibiting to understand instructions or to perform the experimental tasks
* Inability to follow or non-compliance with the procedures of the study
* Contraindications for NIBS or MRI (1):

  * Electronic or ferromagnetic medical implants/device, non-MRI compatible metal implant
  * History of seizures
  * Medication that significantly interacts with NIBS being benzodiazepines, tricyclic antidepressants and antipsychotics
* Regular use of narcotic drugs
* Pregnancy
* Request of not being informed in case of incidental findings
* Concomitant participation in another trial involving probing of neuronal plasticity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Motor learning performance | From baseline to 24 hours after training
  The primary outcome of the study is a laboratory-developed computerized motor task. It is not a standardized clinical scale, but a custom-designed measure specifically created to assess motor learning (e.g., Maceira-Elvira et al. 2022). The task consists of pressing, as quickly and accurately as possible, four buttons corresponding to the fingers labeled from 2 to 5 (2 for the index and 5 for the pinky finger). According to an explicit sequence displayed on a computer screen, the participants learn the sequence. The task performance is evaluated as how fast (sequence, consisting 9 elements/button key presses) and accurate (% of correct sequence) participants perform, within a block of 90 seconds, and their changes over time (during training and following training).

SECONDARY OUTCOMES:
Brain connectivity | Baseline measure (before the intervention)
  Diffusion-weighted and resting-state MRI are performed at baseline, and they allow to evaluate inter-individual anatomical factors associated to the primary outcome. While specific hypotheses exist, particularly regarding cortico-subcortical interactions (i.e., involving striatum), the analyses are exploratory in nature, given complexity of connectivity measures. Functional connectivity will be evaluated using correlation-based methods and graph metrics; structural connectivity will be assessed through diffusion tractography (with graph metrics as well).

CONTACTS AND LOCATIONS:
Locations (2):
- Switzerland (2):
  - EPFL, Campus Biotech, Geneva, Canton of Geneva
  - EPFL Valais, Clinique Romande de readaptation, Sion, Valais

IPD SHARING:
Plan to Share IPD: Undecided